CLINICAL TRIAL: NCT04536350
Title: Inhaled Aviptadil for the Treatment of COVID-19 in Patients at High Risk for ARDS: A Randomized, Placebo Controlled, Multicenter Trial
Brief Title: Inhaled Aviptadil for the Treatment of COVID-19 in Patients at High Risk for ARDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties recruiting participants for the Aviptadil study as there are nowadays very few hospitalized COVID patients. Continuous screening has been carried out but none of the patients met the eligibility criteria for the study.
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Professor of Internal Medicine, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-01902
Record Dates: First submitted 2020-08-21; First posted 2020-09-02 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Covid19; Corona Virus Infection; ARDS; Aviptadil
Keywords: Covid 19; Corona Virus Infection; acute respiratory distress syndrome (ARDS); Aviptadil; Faster recovery
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Distress Syndrome | interventions — aviptadil

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to receive either Aviptadil together with standard care or the placebo (NaCl 0.9%) together with standard care,
Who Masked: Participant, Investigator
Masking Description: Patients and the investigator administering inhalation devices of drug or placebo are not aware of which group they have been randomized to (double-blinded). Someone not involved in the study (e.g. the hospital pharmacist or a nurse not involved in study) prepares the inhalation devices with either drug or placebo according to the randomization plan received by the CTU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aviptadil Treatment (Experimental): Participants will receive standard care plus a dose of 67μg nebulized Aviptadil three times a day for ten days.
  Interventions: Drug: Aviptadil 67μg
- Placebo Treatment (Placebo Comparator): Participants in the control group will receive an Inhalation of 0.9% NaCl solution three times a day for 10 days
  Interventions: Drug: Placebo 0.9% NaCl solution

INTERVENTIONS:
Drug: Aviptadil 67μg — Participants will receive standard care plus a dose of 67μg nebulized Aviptadil three times a day for ten days.
  Arms: Aviptadil Treatment
Drug: Placebo 0.9% NaCl solution — Patiens will receive Standard care plus 0.9% NaCl solution three times a day for ten days
  Arms: Placebo Treatment

SUMMARY:
The world is currently experiencing a coronavirus (CoV-2) pandemic. A new (SARS)-CoV infection epidemic began in Wuhan, Hubei, China, in late 2019; originally called 2019- nCoV the virus is now known as SARSCoV- 2 and the disease it causes COVID-19. Previous CoV epidemics included severe acute respiratory syndrome (SARS)-CoV, which started in China in 2003 and Middle East respiratory syndrome (MERS)-CoV in the Middle East, which started in 2012. The mortality rates were >10% for SARS and >35% for MERS. The direct cause of death is generally due to ensuing severe atypical pneumonia and ensuing acute respiratory distress syndrome (ARDS). Pneumonia also is generally the cause of death for people who develop influenza, although the mortality rate is lower (1%-3% for the influenza A H5N1 pandemic of 1918-1919 in the United States). Risk factors for a poor outcome of SARS-CoV-2 infection have so far been found to include older age and co-morbidities including chronic cardiovascular and respiratory conditions and current smoking status. In May 2020, the FDA authorized the emergency use of remdesivir for treatment of COVID-19 disease based on topline date of two clinical trials, even though an underpowered clinical trial did not find significant improvement in COVID- 19 patients treated with remdesivir. Nevertheless, remdesivir is the first and so far, only approved treatment for COVID-19. Additionally further trials and clinical observations have not found a significant benefit of other antiviral drugs. Although the results of several studies are still pending, there is still a desperate need for an effective, safe treatment for COVID-19. Aviptadil, which is a synthetic form of Human Vasoactive Intestinal Polypeptide (VIP), might be beneficial in patients at risk of developing ARDS. Nonclinical studies demonstrate that VIP is highly concentrated in the lung, where it reduces inflammation.

DETAILED DESCRIPTION:
About 20% of individuals with Corona Virus disease (COVID-19) experience more severe disease characterized by significant respiratory symptoms including acute respiratory distress syndrome (ARDS). ARDS is a known lethal complication due to its low blood oxygenation levels and may result in organ failure. Until now, there are no specific vaccines or therapeutic drugs targeting SARS-CoV-2, alternative therapeutic interventions are needed to prevent and ameliorate respiratory conditions associated with COVID-19 to effectively reduce mortality and prevent ICU admissions. Aviptadil, which is a synthetic form of Human Vasoactive Intestinal Polypeptide (VIP), might be beneficial in patients at risk of developing ARDS. Nonclinical studies demonstrate that VIP is highly concentrated in the lung, where it prevents N-methyl-D-aspartate (NMDA)-induced caspase-3 activation, inhibits IL-6 and TNFa production and protects against HCl-induced pulmonary edema. Further, in animal model systems of lung injury in mice, rats, guinea pigs, sheep, swine and dogs, Aviptadil was shown to restore barrier function at the endothelial/alveolar interface and to protect the lung and other organs from failure. In Europe, Aviptadil is approved for human use and has been shown to be safe in phase II trials for sarcoidosis, pulmonary fibrosis, bronchospasm, erectile dysfunction as well as in a phase I trial in ARDS in the past two decades. In the US, VIP has been given FDA Orphan Drug Designation for the treatment of ARDS and was admitted to the FDA Corona Virus Technology Accelerator Program. In a phase I trial of Aviptadil performed by Sami Said in the early 2000s, eight patients with severe ARDS on mechanical ventilation were treated with ascending doses of intravenous VIP. Seven patients (88%) were successfully extubated and were alive at the five day time point. Six (75%) left the hospital and one (13%) died of an unrelated cardiac event. A phase II clinical trial using intravenous Aviptadil in patients with COVID-19 infection and ARDS has begun. Further, a phase II/III clinical trial will study the effect of inhaled Aviptadil for the treatment of non-acute lung injury in COVID- 19 and begins in June 2020. In Europe, two phase II trials of Aviptadil have been conducted. Further, studies with healthy volunteers have shown that inhaled Aviptadil is well tolerated with few adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection diagnosed
* Risk factors for the development of an ARDS according to an adapted EALI (early acute lung injury score) ≥ 2 Points (with at least one point from the EALI score)

EALI Score:

* 2-6l O2 supplementation to achieve a SaO2>90%: 1 point
* >6l O2 supplementation to achieve a SaO2>90%: 2 points
* Respiratory rate ≥ 30/min: 1 point
* Immunosuppression: 1 Point

Modification (for adapting for risk factors for ARDS in SARS-CoV-2 affected patients

* Arterial hypertension: 1 point
* Diabetes: 1 point
* Fever > 39°C: 1 point

  * Age > 18 years
  * Ability to adequate compliance with the inhalation manoeuvre
  * Ability to sign the informed consent

Exclusion Criteria:

* Known or highly suspected bacterial infection (antibiotic treatment to avoid bacterial superinfection may be allowed)
* PCT ≥ 1μg/l
* Mechanical ventilation
* Inability to conduct inhalation therapy
* Hemodynamic instability with requirement of vasopressor therapy
* Severe comorbidities interfering with the safe participation at the trial according to the treating physician
* Pregnancy
* Systemic immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | Randomization until discharge from hospital but up to maximum 28 days
  Time to clinical improvement of a decrease of at least two points on a seven-point ordinal scale of clinical status or discharged alive from hospital. The seven-point scale consists of the following categories:
  1. not hospitalized;
  2. hospitalized, not requiring supplemental oxygen;
  3. hospitalized, requiring supplemental oxygen;
  4. hospitalized, requiring nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both;
  5. hospitalized, intubation and mechanical ventilation;
  6. ventilation and additional organ support - pressors, renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO);
  7. death

SECONDARY OUTCOMES:
Frequency of mechanical ventilation | Randomization until discharge from hospital up to maximum 28 days
  Frequency of Patient who need mechanical ventilation during hospital stay
Oxygen supplementation | Randomization until discharge from hospital up to maximum 28 days
  Time requiring oxygen supplementation
SaO2 | Randomization until discharge from hospital up to maximum 28 days
  Slope in SaO2
FiO2 | Randomization until discharge from hospital but up to maximum 28 days
  Slope in FiO2
C-reactive Protein | measured at baseline, at least every 7 days and at discharge up to maximum 28 days
  Slope in C-reactive Protein
Neutrophile | measured at baseline, at least every 7 days and at discharge up to maximum 28 days
  Neutrophile ratio
lymphocyte | measured at baseline, at least every 7 days and at discharge up to maximum 28 days
  lymphocyte ratio
Interleukine 6 | measured at baseline, at least every 7 days and at discharge up to maximum 28 days
  Interleukine 6 level
Procalcitonin | measured at baseline, at least every 7 days and at discharge up to maximum 28 days
  Procalcitonin level
Frequency of Multi organ dysfunction Syndrome (MODS) | Randomization until discharge from hospital up to maximum 28 days
  Frequency of Patient who showed a multi organ dysfunction Syndrome during Hospital stay

OTHER OUTCOMES:
Hospitalization | randomization till discharge of hospital up to 28 days
  duration of hospitalization in survivors
treatment initiation to death | Treatment initiation to death up to maximum 28 days
  Time from treatment initiation to death
Blood pressure | Daily until discharge up to maximum 28 days
  Blood pressure will be assessed daily in mmHg
Heart rate | Daily until discharge up to maximum 28 days
  Heart rate will be assessed daily in bpm
Respiratory rate | Daily until discharge up to maximum 28 days
  Respiratory rate will be assessed daily in Counts per minute
Body temperature (auricular) in °C | Daily until discharge up to maximum 28 days
  Body temperature (auricular) will be assessed daily in °C
Pulse oximetry | Daily until discharge up to maximum 28 days
  Pulse oximetry will be assessed daily in %
Glasgow Coma Scale | Daily until discharge up to maximum 28 days
  Glasgow Coma Scale will be assessed daily The lowes possible score is 3 = deep coma or death The highest possible score is 15 = Fully awake
Dispnea and caugh | Randomization until discharge from hospital up to maximum 28 days
  Visual analogue scale for dyspnea and cough as patient-related outcome parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jörg D Leuppi, Professor, Principal Investigator — Cantonal Hosptal, Baselland
Locations (2):
- Switzerland (2):
  - Cantonal Hospital Baselland Liestal, Liestal, Basel-Landschaft
  - Cantonal Hospital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boesing M, Abig K, Brandle M, Brutsche M, Burri E, Frye BC, Giezendanner S, Grutters JC, Haas P, Heisler J, Jaun F, Leuppi-Taegtmeyer AB, Luthi-Corridori G, Muller-Quernheim J, Nuesch R, Pohl W, Rassouli F, Leuppi JD. Inhaled aviptadil for the possible treatment of COVID-19 in patients at high risk for ARDS: study protocol for a randomized, placebo-controlled, and multicenter trial. Trials. 2022 Sep 20;23(1):790. doi: 10.1186/s13063-022-06723-w. PMID 36127739